CLINICAL TRIAL: NCT05789979
Title: The Effectiveness, Feasibility and Potential Risks of Resident Handling Devices in Elderly Residential Setting: A Single Group Pre-post Test Study
Brief Title: The Effectiveness, Feasibility and Potential Risks of Resident Handling Devices in Elderly Residential Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: handling devices_protocol
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Technology
Keywords: Gerontechnology; Resident handling devices; Elderly residential setting

STUDY DESIGN:
Intervention Model Description: The trial is a single group pre-post test study at HOH Nursing Home (NH), Sister Annie Skau Holistic Care Centre (SASHCC), and Care & Attention Home for Severely Disabled (CASD). During the 4-week trial, one floor in SASHCC and one floor in NH will utilize the resident-handling device for residents with high dependency (i.e., lower-limb cannot bear weight). CASD and another floor in NH will use the resident-handling device for residents with low dependency (i.e. lower-limb can bear weight). Outcome indicators are examined during the 1-week pre-test the 4-week trial. Additionally, opinions and comments from care staff and residents regarding the new resident-handling devices will be collected at the end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The resident-handling device (Experimental): This group will use the resident-handling device during the 4-week trial.
  Interventions: Device: The resident-handling device

INTERVENTIONS:
Device: The resident-handling device — Care staff will perform resident-handling tasks using the new resident-handling devices. For low dependency during trial, the device helps care staff to assist residents in making a transition from a sit to a standing posture, vice versa. This device is used for functional activities and transferring and lifting participants. For high dependency during trial, when care staff are performing resident-handling tasks, the device moves with little force in any direction.

SUMMARY:
The study has 12 research questions regarding the use of resident-handling device in elderly residential setting:

Primary study questions:

1. Can the new resident-handling devices improve resident comfortability during the resident-handling task?
2. Are the new resident-handling devices perceived as safe compared to the conventional resident-handling devices?
3. What are the potential risks to the residents and care staff involve in the resident-handling tasks using the new and conventional resident-handling devices?

   Secondary study questions:
4. What are care staff attitudes towards the new and conventional resident-handling devices?
5. What are the perceived difficulties in using the new and conventional resident-handling devices?

   Auxiliary study questions:
6. What are the operation difficulties in the use of the new resident-handling devices in actual operation?
7. What are the perceived benefits and feasibility of using the new resident-handling devices compared to conventional resident-handling devices?
8. [For resident-handling device for residents with low dependency only] Can the new resident-handling device improve resident comfortability in functional activities?
9. [For resident-handling device for residents with low dependency only] Is the new resident-handling device perceived as safe for functional activities compared to the conventional resident-handling devices?
10. [For resident-handling device for residents with low dependency only] What are the potential risks to the residents and care staff involve in functional activities using the new and conventional resident-handling devices?
11. [For resident-handling device for residents with high dependency only] What is the average force exertion of care staff?
12. [For resident-handling device for residents with high dependency only] How frequently does care staff exert excessive force (i.e. Ergo feedback)?

DETAILED DESCRIPTION:
Study design

The trial is a single group pre-post test study at Haven of Hope (HOH) Nursing Home (NH), Sister Annie Skau Holistic Care Centre (SASHCC), and Care & Attention Home for Severely Disabled (CASD). During the 4-week trial, one floor in SASHCC and one floor in NH will utilize the resident-handling device for residents with high dependency (i.e., lower-limb cannot bear weight). CASD and another floor in NH will use the resident-handling device for residents with low dependency (i.e. lower-limb can bear weight). Outcome indicators are examined during the 1-week pre-test the 4-week trial. Additionally, opinions and comments from care staff and residents regarding the new resident-handling devices will be collected at the end of the trial.

This protocol complies with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Guideline for Good Clinical Practice (ICH-GCP) and Declaration of Helsinki.

Subjects

1. Residents

   Residents of two selected floors at Nursing Home (NH), Care & Attention for Severely Disabled (CASD), and Sister Annie Skau Holistic Care Centre (SASHCC) will be recruited.

   Inclusion criteria for high dependency device:

   • Lower limb cannot bear weight,
   * Assessed by health care workers (e.g., occupational therapists, physiotherapists, nurses) that manual handling is not appropriate
   * According to the study site instruction, require the use of resident handling device

   Exclusion criteria:
   * None

   Inclusion criteria for low dependency device:

   • Lower-limb can bear weight

   • Assessed by health care workers (e.g., occupational therapists, physiotherapists, nurses) that manual handling is not appropriate

   • According to the study site instruction, require the use of resident handling device

   Exclusion criteria:

   • None
2. Care staff Care staff of two selected floors at Nursing Home (NH), Care & Attention for Severely Disabled (CASD), and Sister Annie Skau Holistic Care Centre (SASHCC) will be recruited.

Inclusion criteria:

• Responsible for transferring and lifting residents using any of the new resident handling devices

Exclusion criteria:

• None

Procedures

1. Participants' recruitment and consent

   The criteria stated in the Alzheimer Europe Report (2011) will be followed to ensure that the participants are provided chances to give consent. In particular, four criteria will be evaluated, including 1) the person must have sufficient capacity to understand the information, 2) the person is able to retain, use and weight up such information for making a decision, 3) the person will understand the benefit, risk, and convenience, 4) the person must have the ability to communicate the decision. The University of Hong Kong (HKU) research staff and the care staff will first commit them in a causal chat to assess their ability to communicate and understand the dialogues. If residents meet all the four criteria, both residents and their next of kin will be approached for consent. Otherwise, only their next of kin will be approached for consent.

   For the residents who will be approached for consent, the HKU research staff will elaborate the study based on the opt-out consent script and give them the opt-out consent document. Neither HKU nor the supplier will get personal or sensitive information of the participants due to the study. If they do not want to participate, they can notify the care staff. Unless they indicate withdrawal from the study, they are treated as consenting to join the study (opt-out participation). Every time before using the devices, the care staff will inform the use of the devices. Devices will be used only when participants do not raise objections.

   Their next of kin will be informed of the new devices and the study through standard channel of the test site (i.e. messaging mobile phone app or phone). If they do not want the residents to participate, they can notify the care staff. Unless they indicate withdrawal from the study, they are treated as consenting the residents to join the study (opt-out participation).

   For the care staff, it will be presumed that they agree to participate in the study if they complete the anonymous questionnaire (implied consent).

   Before qualitative interviews with the participants, written consent will be obtained from them and their next of kin. Before qualitative interviews with the care staff, written consent will be obtained from them.
2. Baseline data collection

   Before the trial, all test sites use the conventional resident-handling devices available in their service units. In the week before the trial, the baseline data of the level of comfort during transfer and lifting, care staff attitudes towards the conventional resident-handling devices and perceived difficulties in using conventional resident-handling devices will be collected. It is a standard practice for the study site to require all staff operating the devices to pass yearly audit to ensure that they can operate the devices properly. Potential risks to residents and care staff during using the conventional resident-handling device resident-handling and/or functional activities will be assessed based on the audit reports in last year. The safety audit reports will be provided by study site manager.
3. Training of resident-handling device for care staff

   A few 1.5- to 2-hour trainings on the use of resident-handling device will be delivered to all care staff. During the training, care staff will learn how to use the device with hands-on experience. Also, the product supplier will provide a 10-minute demonstration video for care staff to better understand the operation procedure. A protocol detailing related device operations will be prepared for the staff.
4. Safety audit

   After the staff training, care staff who are responsible for transferring and lifting residents using the new resident-handling devices will be audited by clinical professionals (e.g., occupational therapists, physiologists) to ensure that they can operate the devices properly. The audit items are developed based on the experience of using and auditing various types and models of resident-handling devices of the study sites, and are in use for years. The audit takes around 2 to 3 weeks to complete. Potential risks to residents and care staff during using the new resident-handling device for resident-handling and/or functional activities will be assessed based on the audit reports. The safety audit reports will be provided by study site manager.
5. Implementation

   Care staff at one selected floor of Nursing Home (NH) and Care & Attention for Severely Disabled (CASD) will use the resident handling device for participants with low dependency during the 4-week trial. The device helps care staff to assist residents in making a transition from a sit to a standing posture, vice versa. This device is used for functional activities and transferring and lifting participants.

   On the other hand, care staff at another selected floor at Nursing Home (NH) and Sister Annie Skau Holistic Care Centre (SASHCC) will use the resident handling device for residents with high dependency during the 4-week trial. When care staff are performing resident handling tasks, the device moves with little force in any direction. The handlebar's force sensors detect and transfer force in the appropriate directions, speeding up the 5th wheel below. There will be a real-time alert if the care staff pushes or pulls at a force more than 20 kilogram (which should not be exceeded as per the recommendation of Occupational Safety and Health Council).
6. Trial data collection

In the first trial week, clinical consultant(s) will observe the actual operation for once for each device model to investigate operation difficulties, and record the observations in an observation report. Operation protocol may be revised. A 5 to 15 minutes follow-up staff training may be delivered to all care staff based on the revised protocol.

During the 4-week trial, care staff will complete a self-administrated questionnaire about the level of comfort expressed by residents and perceived safety when they perform resident handling and/or functional activities using the resident handling device every week.

At the end of the trial, 2 to 4 residents and 3 to 4 cares staff at each test site will be selected by convenience and invited to an interview. Interview contents include the perceived benefits and feasibility of new resident handling devices compared to conventional resident handling devices. For the resident handling device for participants with high dependency, data of care staff's average force exertion and number of Ergo feedback (a proxy measure of number of times care staff use excessive force) will be retrieved.

Blinding

No blinding will be done for this single group study.

Sample size determination

The sample size is estimated by the current number of care staff who are responsible for resident handling tasks and residents who require the use of resident handling device at the study sites. It is estimated that a total of 35 residents and 28 care staff will be using the resident handling device for residents with high dependency, while a total of 22 residents and 35 care staff will be using the resident handling device for residents with low dependency.

Data analysis

1. Main analysis

   Independent sample t-test will be used to evaluate the change in the anonymous pre-post data of level of comfort expressed by residents, perceived safety, care staff attitudes towards the resident-handling device and perceived difficulties in using of new resident-handling device. Independent sample t-test with Bonferroni correction will be used to evaluate the change in the anonymous weekly data of level of comfort expressed by residents, perceived safety, care staff attitudes towards the resident-handling device and perceived difficulties in using of new resident-handling device.

   Safety audit reports regarding the potential risks involved in the resident-handling tasks and functional activities during pre-test and trial period will be compared.

   Descriptive statistics will used to show the average force that care staff exert and number of Ergo feedback (a proxy measure of number of times care staff use excessive force) generated by the device.

   The operation difficulties in the use of the new resident-handling devices in actual operation will be summarised.
2. Qualitative interview

The content will be transcribed verbatim in Chinese for further analysis. Transcripts will be analysed using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the new and conventional resident-handling device. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for high dependency device:

* Lower limb cannot bear weight,
* Assessed by health care workers (e.g., occupational therapists, physiotherapists, nurses) that manual handling is not appropriate
* According to the study site instruction, require the use of resident-handling device

Inclusion criteria for low dependency device:

* Lower-limb can bear weight
* Assessed by health care workers (e.g., occupational therapists, physiotherapists, nurses) that manual handling is not appropriate
* According to the study site instruction, require the use of resident-handling device

Inclusion criteria for care staff:

• Responsible for transferring and lifting residents using any of the new resident-handling devices

Exclusion Criteria:

Exclusion criteria for high dependency device, low dependency device and care staff:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
5-week change in the level of comfort expressed by residents | From the start of 1-week pre-test to the end of the 4-week trial period
  Care staff will complete an item indicating the level of comfort expressed by residents in using the conventional and new resident handling devices on a 5-point Likert scale (i.e. 1 indicating very uncomfortable and 5 indicating very comfortable). The minimum and maximum values of the scale are 1 and 5 respectively. Higher score indicates higher level of comfort.
5-week change in perceived safety | From the start of 1-week pre-test to the end of the 4-week trial period
  Care staff will complete two items indicating the perceived safety in using the conventional and new resident handling devices on a 5-point Likert scale (i.e. 1 indicating very unsafety and 5 indicating very safety). The minimum and maximum values of the scale are 2 and 10 respectively, with higher score indicating higher level of safety.
Qualitative measures: The potential risks to residents and staff involved in resident-handling tasks | Within a year before the 4-week trial to before the start of the 4-week trial
  Potential risks to residents and care staff during the use of the new resident handling device for resident handling and/or functional activities will be assessed based on the audit reports. The safety audit reports will be provided by study site manager. Safety audit reports regarding the potential risks involved in the resident-handling tasks and functional activities during pre-test and trial period will be compared. The contents include the preparation of residents and environment, the preparation of staff and tools, the operation process and the aftermath.

SECONDARY OUTCOMES:
Care staff attitudes towards resident-handling devices | From the start of 1-week pre-test to the end of the 4-week trial period
  Care staff will complete four items indicating their attitudes towards conventional and new resident handling devices in the past week at week 0 and 4 on a 5-point Likert scale (i.e. 1 indicating strongly disagree and 5 indicating strongly agree). The minimum and maximum values of the scale are 4 and 20 respectively, with higher score indicating higher level of acceptability.
Perceived easiness in using resident-handling devices | From the start of 1-week pre-test to the end of the 4-week trial period
  Care staff will complete nine items indicating the perceived easiness in using conventional and new resident handling devices on a 5-point Likert scale (i.e. 1 indicating many difficulties and 5 indicating no difficulties) in the past week at week 0 and 4. The minimum and maximum values of the scale are 8 and 40 respectively, with higher score indicating perceived easier use of the devices.
Qualitative measures: The operation difficulties in the use of the new resident-handling devices in actual operation | In the first week of the 4-week trial period
  In the first trial week, clinical consultant will observe the actual operation for once for each device model to investigate operation difficulties and record the observation in an observation report.
Qualitative measures: The perceived benefits and feasibility of the resident-handling devices of residents | At the end of the 4-week trial period
  At the end of the trial, 2 to 4 residents at each test site will be selected by convenience and invited to an interview. Interview contents include the perceived benefits and feasibility of new resident-handling devices compared to conventional resident-handling devices.
  1. Is it safe in using the new handling devices during transfer and lifting and/or functional activities?
  2. Do you feel comfortable in using new handling devices during transfer and lifting and/or functional activities?
  3. On the whole, are you satisfied with the new handling devices?
  4. Do you want the service unit to continue to use the new handling devices in the future?
Qualitative measures: The perceived benefits and feasibility of the resident-handling devices of care staff | At the end of the 4-week trial period
  At the end of the trial, 3 to 4 cares staff at each test site will be selected by convenience and invited to an interview. Interview contents include the perceived benefits and feasibility of new resident-handling devices compared to conventional resident-handling devices.
  1. Do you want bigger or smaller size of handling devices?
  2. Is the new handling device safe?
  3. Is there any abnormal operation during the testing?
  4. Is there any accident during the testing?
  5. What can be improved in using the new handling devices?
  6. Is it easy to operate?
  7. Does it spend less time in operation?
  8. What is the attitude of residents?
  9. Do the new handling devices fulfill your expectation?
  10. Can you give advice to other care staff while using this handling device?
  11. Do you worry about using the new handling devices or refuse to use because of wrong operation?
The level of comfort expressed by residents with low dependency on using the functional activities | From the start of 1-week pre-test to the end of the 4-week trial period
  Care staff will complete an item indicating the level of comfort expressed by residents with low dependency in using new resident handling devices on a 5-point Likert scale (i.e. 1 indicating very uncomfortable and 5 indicating very comfortable). The minimum and maximum values of the scale are 1 and 5 respectively. Higher score indicates higher level of comfort.
Perceived safety of residents with low dependency on using the functional activities | From the start of 1-week pre-test to the end of the 4-week trial period
  Care staff will complete two items indicating the perceived safety on using the functional activities of new handling devices on a 5-point Likert scale (i.e. 1 indicating very unsafety and 5 indicating very safety). The minimum and maximum values of the scale are 2 and 10 respectively, with higher score indicating high level of safety.
Qualitative measures: The potential risks to residents with low dependency and staff when the device is used for functional activities | Within a year before the 4-week trial to before the start of the 4-week trial
  Potential risks to residents and care staff during the use of the new resident handling device for resident handling and/or functional activities will be assessed based on the audit reports. The safety audit reports will be provided by study site manager. Safety audit reports regarding the potential risks involved in the resident-handling tasks and functional activities during pre-test and trial period will be compared. The contents include the preparation of residents and environment, the preparation of staff and tools, the operation process and the aftermath.
The average force exertion of care staff on residents with high dependency | From the start to the end of the 4-week trial period
  The average force that care staff exert in using the high dependency device will be generated by the device.
The number of Ergo feedback (a proxy measure of the number of times care staff use excessive force) of residents with high dependency | From the start to the end of the 4-week trial period
  The number of Ergo feedback (a proxy measure of number of times care staff use excessive force) will be generated by the device.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Haven of Hope Hang Hau Care and Attention Home for Severely Disabled, Hong Kong
  - Haven of Hope Nursing Home, Hong Kong
  - Haven of Hope Sister Annie Skau Holistic Care Centre, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.